CLINICAL TRIAL: NCT04354896
Title: The Effect of Thyroid Hormone Therapy on Muscle Mass and Function in Older Adults With Subclinical Hypothyroidism - a Substudy of TRUST and IEMO Trials
Brief Title: The Effect of Thyroid Hormone Therapy on Muscle Mass and Function in Older Adults With Subclinical Hypothyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 320030_172676; 2011-004554-26 (EudraCT Number); 2012-004160-22 (EudraCT Number)
Record Dates: First submitted 2020-04-08; First posted 2020-04-21 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Subclinical Hypothyroidism; Sarcopenia
Keywords: Physical performance; muscle mass; muscle function
MeSH Terms: conditions — Sarcopenia | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levothyroxine (Experimental): The intervention will start with Levothyroxine 50 mcg daily with regular blinded dosis titration.
  Interventions: Drug: Levothyroxin
- Placebo (Placebo Comparator): Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxin — The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH 0.4 to 4.6 mU/L, no change to dose; TSH ≥4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Arms: Levothyroxine
Drug: Placebo — Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug.
  Arms: Placebo

SUMMARY:
Subclinical hypothyroidism (SCH) is common among the elderly population and has been associated with neuromuscular impairment. Muscular symptoms such as weakness, myalgia and cramps are more often reported by SCH patients compared to euthyroid controls. Sarcopenia is the age-related loss of muscular mass and function and its assessment includes three dimensions (muscle quantity, muscle strength and physical performance). To date, evidence is lacking about the effect of thyroid hormone replacement on skeletal muscle impairment in SCH patients. The aim of the study is therefore to evaluate the impact of levothyroxine therapy on sarcopenia measures in SCH. This is a nested substudy within two large international multicenter randomized controlled trial of elderly participants with SCH (TRUST Study, clinicaltrials.gov ID NCT 01660126; and IEMO Study, Netherland Trial Register ID NTR3851). Those two trials shared a very similar study design. The cohorts will therefore be analyzed as a single study population.

DETAILED DESCRIPTION:
Background

Subclinical hypothyroidism (SCH) is common among the elderly population, with an estimated prevalence of 6-15%. It has been associated with multiple adverse outcomes such as cardiovascular diseases and neuropsychological disturbance. Muscular function impairment has also been associated with SCH. However, the association between subclinical hypothyroidism and physical performance in older adults remains unclear and randomized controlled trials are lacking.

Physical performance is an important prognostic indicator for older adults. Prospective studies showed that it is related to hospitalization, institutionalization, cardiovascular disease, disability and mortality. Gait speed is one of the most widely used measures of physical performance in clinical and research settings, with a solid prognostic value.

Aside from overall physical performance, two other dimensions of muscular function can be assessed: muscle function, usually assessed by handgrip strength (predictive validity for decline in cognition, mobility, functional status and mortality for older people), and muscle mass, usually assessed by dual-energy X-absorptiometry). Those three dimension together form the definition of sarcopenia, a relatively new concept which has been gaining visibility in the last years because of its high prevalence and clinical relevance.

Both subclinical hypothyroidism and muscle function impairment are highly prevalent among the older population, and the latter bears a heavy personal, social and economic burden. Therefore, evaluating the potential benefit of levothyroxine therapy on muscle function in this population holds the potential to prevent adverse health-related outcomes and maintain the patients' autonomy and quality of life.

Objectives

To investigate whether levothyroxine therapy in older adults with subclinical hypothyroidism affects sarcopenia measures (mass, strength and physical performance) in a substudy of the TRUST and IEMO trial.

Methods

The existing trial infrastructure (TRUST and IEMO trials, clinicaltrials.gov ID: NCT 01660126) will be utilized to collect information on muscle mass and function from 322 participants with persistent subclinical hypothyroidism randomized to either thyroxine or placebo. Utilized outcomes are specified in the corresponding section.

ELIGIBILITY:
Inclusion Criteria (TRUST):

* Community-dwelling elderly patients aged ≥65 years with subclinical hypothyroidism (SCH).

[SCH is defined as elevated TSH levels (4.6 to 19.9 mU/L) and free thyroxine (fT4) in reference range measured on a minimum of two occasions at least 3 months apart.]

Inclusion Criteria (IEMO)

- Community-dwelling elderly patients aged ≥80 years with SCH, as above defined

Exclusion Criteria (TRUST and IEMO):

* Currently on Levothyroxine or antithyroid drugs, amiodarone or lithium.
* Recent thyroid surgery or radio-iodine (within 12 months).
* Grade IV NYHA heart failure.
* Prior clinical diagnosis of dementia.
* Recent hospitalisation for major illness or elective surgery (within 4 weeks).
* Recent acute coronary syndrome, including myocardial infarction or unstable angina (within 4 weeks).
* Terminal illness.
* Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Individuals participating in ongoing RCTs of therapeutic interventions (including CTIMPs)
* Individuals planning to move out of the region in which the trial is being conducted within the next 2 years (proposed minimum follow-up period).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 322 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Physical performance | Final visit (12 to 42 months after baseline visit)
  Gait speed (3-meter and 6-meter walk test) [m/s]

SECONDARY OUTCOMES:
Muscle mass | Baseline, 1-year follow up and/or 2-year follow-up (yearly change)
  ALM/BMI, i.e. appendicular lean mass (ALM) assessed with Dual-Energy X-Ray Absorptiometry [kg], divided by body mass index [kg/m2]
Muscle strength | Baseline, 1-year follow-up
  Handgrip strength, measured with a Jamar isometric Dynamometer [kg]
Sarcopenia | Final visit (12 to 42 months after baseline visit)
  Sarcopenia diagnostic criteria are applied to each participant with all three Outcomes (gait speed, handgrip strength, DXA) at the end of follow-up. E.g., a participant is diagnosed with sarcopenia when muscle mass measured with DXA is decreased (ALM/BMI for men < 0.79, for women < 0.51), in the presence of impaired grip strength (for men <27 kg, for women <16 kg). If present, sarcopenia is further classified as "severe" in presence of a gait speed<0.8 m/s.
  The proportion of sarcopenic individuals between the levothyroxine and the placebo groups is then compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD MAS, Principal Investigator — BIHAM UniBern
Locations (5):
- Netherlands (3):
  - Department of Gerontology and Geriatrics, Leiden University Medical Center, Leiden
  - Department of Public Health and Primary Care, Leiden University Medical Center, Leiden
  - Institute for Evidence-Based Medicine in Old Age, Leiden
- Switzerland (2):
  - Department of General Internal Medicine, Lausanne, Canton of Vaud
  - Clinic for General Internal Medicine, Bern University Hospital Bern, Bern

REFERENCES:
- [Background] Stott DJ, Rodondi N, Kearney PM, Ford I, Westendorp RGJ, Mooijaart SP, Sattar N, Aubert CE, Aujesky D, Bauer DC, Baumgartner C, Blum MR, Browne JP, Byrne S, Collet TH, Dekkers OM, den Elzen WPJ, Du Puy RS, Ellis G, Feller M, Floriani C, Hendry K, Hurley C, Jukema JW, Kean S, Kelly M, Krebs D, Langhorne P, McCarthy G, McCarthy V, McConnachie A, McDade M, Messow M, O'Flynn A, O'Riordan D, Poortvliet RKE, Quinn TJ, Russell A, Sinnott C, Smit JWA, Van Dorland HA, Walsh KA, Walsh EK, Watt T, Wilson R, Gussekloo J; TRUST Study Group. Thyroid Hormone Therapy for Older Adults with Subclinical Hypothyroidism. N Engl J Med. 2017 Jun 29;376(26):2534-2544. doi: 10.1056/NEJMoa1603825. Epub 2017 Apr 3. PMID 28402245
- [Background] Stott DJ, Gussekloo J, Kearney PM, Rodondi N, Westendorp RG, Mooijaart S, Kean S, Quinn TJ, Sattar N, Hendry K, Du Puy R, Den Elzen WP, Poortvliet RK, Smit JW, Jukema JW, Dekkers OM, Blum M, Collet TH, McCarthy V, Hurley C, Byrne S, Browne J, Watt T, Bauer D, Ford I. Study protocol; Thyroid hormone Replacement for Untreated older adults with Subclinical hypothyroidism - a randomised placebo controlled Trial (TRUST). BMC Endocr Disord. 2017 Feb 3;17(1):6. doi: 10.1186/s12902-017-0156-8. PMID 28158982
- [Background] Mooijaart SP, Du Puy RS, Stott DJ, Kearney PM, Rodondi N, Westendorp RGJ, den Elzen WPJ, Postmus I, Poortvliet RKE, van Heemst D, van Munster BC, Peeters RP, Ford I, Kean S, Messow CM, Blum MR, Collet TH, Watt T, Dekkers OM, Jukema JW, Smit JWA, Langhorne P, Gussekloo J. Association Between Levothyroxine Treatment and Thyroid-Related Symptoms Among Adults Aged 80 Years and Older With Subclinical Hypothyroidism. JAMA. 2019 Nov 26;322(20):1977-1986. doi: 10.1001/jama.2019.17274. PMID 31664429
- [Derived] Netzer S, Chocano-Bedoya P, Feller M, Janett-Pellegri C, Wildisen L, Buchi AE, Moutzouri E, Gonzalez Rodriguez E, Collet TH, Poortvliet RKE, Mc Carthy VJC, Aeberli D, Aujesky D, Westendorp R, Quinn TJ, Gussekloo J, Kearney PM, Mooijaart S, Bauer DC, Rodondi N. The effect of thyroid hormone therapy on muscle function, strength and mass in older adults with subclinical hypothyroidism-an ancillary study within two randomized placebo controlled trials. Age Ageing. 2023 Jan 8;52(1):afac326. doi: 10.1093/ageing/afac326. PMID 36721961